CLINICAL TRIAL: NCT03241290
Title: Prospective Assessment of the Quality of the Image and the Usability of the C-ARM ARCO FP-Rk521S Used in Surgical Conventional Practice
Brief Title: Assessement of the C-ARM ARCO FP-Rk521 S in Surgical Conventional Practice
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Clinical Investigation Centre for Innovative Technology Network (Network)
Responsible Party: Sponsor
Other Study IDs: 38RC17.010; 2017-A00103-50 (Other: ID RCB)
Record Dates: First submitted 2017-07-03; First posted 2017-08-07 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: C.Surgical Procedure
Keywords: C-arm; Medical Imaging Device; Radiological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Use of C-ARM ARCO FP-Rk521S: C-ARM ARCO FP-Rk521S is mobile X-ray device that combines a X-Ray sensor and a sensor management software used during surgeries for real-time imaging.

SUMMARY:
THALES-EVAQUAL study assesses the quality of the images generated by C-ARM ARCO FP-Rk521S and its ability to be used during surgery.

DETAILED DESCRIPTION:
Expected performance of TED developped technology compared to current equipment (intensifier tube) represent a significant improvement; especially in term of image rendering, irradiation dose reduction and ergonomy.

THALES-EVAQUAL is a prospective,monocentric, unrandomized, and uncontrolled study which objective is to assess C-ARM ARCO FP-Rk521S in term of quality of image. It also evaluates its ability to be used during Orthopedic, neurological and neurological surgeries.

Patient included in the study will have a surgery during which C-ARM is used. This study doesn't modify the medical care of the patient.

After each surgery, a digital scale of image quality will be filled by the surgeon for each aquisition. Other feedback questionnaires regarding the suitability of the device and the satisfaction of the surgeon will also be completed.

ELIGIBILITY:
Inclusion Criteria:

* Subject having signed the non-objection form;
* Requiring one of the following surgical procedures:

  * Urology: soft ureteroscopy, uteroscopy, sacral neuromodulation, JJ sent placement.
  * Orthopedics: vertebroplasty, gamma nail placement, sacro-iliac screw fixation.
  * Neurology: spinal surgery

Exclusion Criteria:

* Subject who refuse to participate in the study;
* Who are under legal protection measure or unable to express their consent (guardianship, curatorship);
* Deprived of liberty by judicial or administrative decision.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who undergo surgery (orthopedic, urological or neurological surgery)
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2017-05-29 (Actual); Primary Completion 2018-12-11 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
Digital scale of image quality | up to 5 hours
  Digital scale of image quality completed for each acquisition by the surgeon

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Moreau-Gaudry, MD, PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital, Grenoble, Grenoble, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Clinical Investigation Centre for Innovative Technology Network website — http://www.cic-it.fr/cic-it-grenoble.php